CLINICAL TRIAL: NCT01626950
Title: Living Conditions and Breast Cancer
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AO/INCA/2011/JPD; 2012-A00377-36 (Other: ANSM)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-03

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; living conditions; social fragility
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases - Stage III-IV breast cancer: The women in this group have been diagnosed with stage III-IV incident cancer.
- Controls: Stage I-II breast cancer: The women in this group have been diagnosed with stage I-II incident cancer.

SUMMARY:
The main objective of this study is to estimate of the link (odds ratio) between the precariousness defined by the score SPICE (2 groups: precarious and insecure) and stage at diagnosis (2 groups: CAS: stages 1 or 2 the "good prognosis "versus the witnesses: stage 3 or 4 bad prognosis).

DETAILED DESCRIPTION:
Our secondary objectives include:

* To study the link between cancer stage at diagnosis and diverse parameters describing living conditions
* To construct a new score for social fragility based on new data collected in this study, and to compare this score with the EPICES score
* To study patient quality of life at study baseline

ELIGIBILITY:
Inclusion Criteria (for cases):

* Patient has been correctly informed about the study, and agrees to participate
* The patient must be insured or beneficiary of a health insurance plan
* Incident breast cancer cases (diagnosis based on pathology) excluding sarcoma, classifiable as stage III-IV, surgical cases

Inclusion Criteria (for controls):

* Patient has been correctly informed about the study, and agrees to participate
* The patient must be insured or beneficiary of a health insurance plan
* Incident breast cancer cases (diagnosis based on pathology) excluding sarcoma, classifiable as stage I-II, surgical cases

Exclusion Criteria (for cases and controls):

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient is pregnant, parturient, or breastfeeding
* The patient is opposed to study participation
* Women not able to answer a questionnaire due to language barriers or due to vascular or degenerative cerebral dysfunction
* It is impossible to correctly inform the patient

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a case-control study concerning the female population suffering from breast cancer in the Herault department of France. Only invasive cancers are taken into account. For each case, we will have at least 2 controls, matched according to age +- 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11-18 (Actual); Study Completion 2013-11-18 (Actual)

PRIMARY OUTCOMES:
The odds ratio for having a stage I-II diagnosis versus a stage III-IV diagnosis according to EPICE score category (social fragility versus no social fragility). | Baseline (Day 0; cross-sectional study)
  The main criterion is the estimation of the link (odds ratio) between the precariousness defined by the score SPICE (2 groups: precarious and insecure) and stage at diagnosis (2 groups: CAS: stages 1 or 2 the "good prognosis "versus the witnesses: stage 3 or 4 bad prognosis).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre Daurès, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - IURC - Laboratoire de Biostatistique d'Epidémiologie et de Recherche Clinique, Montpellier
  - Equipe Démographie Santé, Montpellier
  - Registre Tumeurs de l'Hérault, Montpellier

REFERENCES:
- [Result] Orsini M, Tretarre B, Daures JP, Bessaoud F. Individual socioeconomic status and breast cancer diagnostic stages: a French case-control study. Eur J Public Health. 2016 Jun;26(3):445-50. doi: 10.1093/eurpub/ckv233. Epub 2016 Jan 28. PMID 26823441